CLINICAL TRIAL: NCT04797468
Title: A Phase 1 Clinical Study to Investigate the Safety, Tolerability and to Determine the Maximum Tolerated Dose and Recommended Phase 2 Dose of HLX23 (CD73 Inhibitor) in Patients With Advanced or Metastatic Solid Tumors
Brief Title: A Phase 1 Study of the CD73 Inhibitor(HLX23) Alone in Participants With Solid Tumor
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The Early Termination is the result of the sponsor's need to reevaluate the study design and to make needed vendor realignments.
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HLX23-001
Record Dates: First submitted 2021-03-04; First posted 2021-03-15 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HLX23 (Experimental): HLX23 administered IV.
  Interventions: Drug: HLX23

INTERVENTIONS:
Drug: HLX23 — administered IV.
  Other Names: CD73 inhibitor

SUMMARY:
The reason for this study is to see if the CD73 inhibitor HLX23 alone is safe and effective in participants with advanced solid cancer.

DETAILED DESCRIPTION:
An open-label, dose escalation, first-in-human, phase 1 clinical study to investigate the safety, tolerability and to determine the maximum tolerated dose and recommended phase 2 dose of HLX23 (recombinant anti-CD73 humanized monoclonal antibody) in patients with advanced or metastatic solid tumors

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate, fully understand the study and have signed the ICF, willing and have the capacity to comply with and complete all trial procedures;
2. Aged ≥ 18 years when signing the ICF;
3. Patients with advanced or metastatic solid tumors confirmed by histologically or cytologically, who have failed standard treatment, or who do not have standard treatment regimens, or who are not suitable for standard treatment;
4. Patients with at least one evaluable lesion assessed as per RECIST1.1 criteria;
5. Patients must be able to supply adequate tumor tissue for biomarker (CD73 and CD68 ) analyses;
6. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 when enrolled in the study;
7. Life expectancy longer than three months;
8. Adequate hematologic functions;
9. Adequate hepatic function ;
10. Adequate renal function, as defined by the creatinine clearance rate ≥ 50 mL/minute by Cockcroft-Gault formula;
11. Adequate cardiac function ;
12. At least 28 days from prior major surgery or medical device or local radiotherapy, at least five half-lives from prior cytotoxic chemotherapy, immunotherapy, biological agents and at least 14 days from prior hormonal therapy and minor surgery before the first infusion of HLX23;
13. For patients with hepatocellular carcinoma, the Child-Pugh score has to be A;
14. Female participants of childbearing potential and male partners with female partners of childbearing potential must agree to use one adequate and medically approved barrier method of contraception during the study and for at least 6 months after the last dose of the study drugs.

Exclusion criteria:

1. Patients who still have ≥ grade 2 toxicities from prior therapies;
2. Patients who have history of allergic reaction to monoclonal antibodies;
3. Concurrent unstable or uncontrolled medical conditions;
4. Any concurrent malignancy other than basal cell carcinoma or carcinoma in situ of the cervix (patients with previous history of malignancy but without evidence of disease for ≥ 3 years can participate in the study);
5. History of prior treatment with anti-CD73 antibodies,including patients treated with adenosine receptor antagonists, CD39 or CD73 inhibitors ;
6. Patients with active autoimmune disease, except vitiligo or cured childhood asthma/allergies that requires no intervention after adulthood, autoimmune-mediated hypothyroidism treated with stable doses of thyroid hormone replacement, or Type I diabetes treated with stable doses of insulin can be excepted. Patients in a stable state and do not require systemic immunosuppressive therapy (including corticosteroids) are allowed to be enrolled;
7. Pregnancy or breast-feeding;
8. Known history of human immunodeficiency virus infection (HIV), but the patients with CD4+ T-cell (CD4+) counts ≥ 350 cells/uL are allowed to be enrolled.
9. hepatitis B virus carrier status (HBV surface antigen positive) and hepatitis C carrier (anti-HCV antibody positive). If HBsAg (+) or HBcAb (+), the HBV-DNA≥2500copy/mL or 500 IU/mL, or clinically judged active hepatitis; Subjects co-infected with hepatitis B and hepatitis C should be excluded (positive HBsAg or HBcAb test and positive HCV antibody test);
10. The patient is the investigator, sub-investigator or anyone directly involved in the conduct of the study;
11. History or current evidence of any condition or disease that could confound the results of the study, or participation is not in the best interest of the patient in the opinion of the Investigator(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Dose Limiting Toxicity | Up to 21 Days
  DLT
maximum tolerated dose of HLX23 | Up to 21 Days
  MTD
Recommended phase 2 dose of HLX23 | Up to 21 Days
  RP2D

SECONDARY OUTCOMES:
Pharmacokinetics(PK) | cycle 1 (one week is a cycle) to day 30 after the last dose
  To measure the serum concentration of HLX23
Pharmacodynamic(PD) | cycle 1, cycle 2, cycle 3 (one week is a cycle) to day 30 after the last dose
  Percentage of CD73 receptor occupancy on circulating
Immunogenicity | cycle 1, cycle 2, cycle 4, cycle 6 to day 30 after the last dose
  Incidence of anti-HLX23 antibody (ADA) positive results
Overall Response Rate (ORR) | Baseline through Disease Progression or Death (Estimated at up to 2 Years)
  Percentage of Participants with Complete Response (CR) or Partial Response (PR)
Disease Control Rate (DCR) | Baseline through Measured Progressive Disease (Estimated at up to 2 Years)
  Percentage of Participants with a Best Overall Response of CR, PR, and Stable Disease

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Research Site, Los Angeles, California
  - Research Site, Orange, California
  - Research Site, Orange City, Florida
  - Research Site, Fairway, Kansas
  - Research Site, Detroit, Michigan
  - Research Site, Greenville, South Carolina